CLINICAL TRIAL: NCT05190146
Title: A Multi-country, Epidemiologic Study to Assess the Interferon Gamma Release Assay (IGRA) Positivity, and to Build Capacity to Conduct a Tuberculosis (TB) Vaccine Efficacy Study, in Populations With a High TB Disease Burden
Brief Title: Epidemiologic Study to Assess the IGRA Positivity in Populations With a High TB Burden
Status: Completed | Type: Observational
Sponsor: Gates Medical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Gates MRI TBV02-E01
Record Dates: First submitted 2021-11-29; First posted 2022-01-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for primary, secondary and exploratory endpoints; sputum samples for secondary and exploratory endpoints; and urine sample for exploratory endpoints
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to conduct a multi-country, multi-site, epidemiologic study designed to assess the proportion of interferon gamma release assay (IGRA) positivity, at site level, and to build capacity to conduct a future TB vaccine efficacy study.

ELIGIBILITY:
Inclusion Criteria: Capable of giving signed informed consent and informed assent (as appropriate), which includes compliance with the requirements listed in the informed consent form (ICF) and informed assent form (IAF)

Between 15 and 34 years of age (inclusive)

Participants who agree to stay in contact with the study site for the duration of the study, provide updated contact information as necessary, and have no current plans to relocate from the study area for the duration of the study.

Exclusion Criteria:

History of active TB within the last 24 months (i.e., 24 months from end of treatment to day of screening, based on history [no documentation required])

History of previous administration of an experimental Mtb vaccine

Unstable / uncontrolled chronic condition according to the judgment of the investigator

-

Ages: 15 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A maximum of 7,203 participants who are at high risk of Mtb infection and TB (disease) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 7203 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
IGRA status per site | Screening
  Proportion of participants with a positive IGRA, per site, calculated using per protocol population. 95% CI will summarize the precision associated with the estimate.

SECONDARY OUTCOMES:
IGRA status by age group per site | Screening
  Proportion of participants with a positive IGRA, by age group (15 to 24 [inclusive], and 25 to 34 years of age [inclusive]) per site, calculated using per protocol population. 95% CI to summarize the precision associated with the estimates.
Suspected pulmonary TB during follow-up period | Day 1 up to 30 months
  Incidence rate of participants with suspected TB to be summarized by country. Exact 95% CI to be provided
Laboratory-confirmed pulmonary TB during follow-up period | Day 1 up to 30 months
  Incidence rate of participants with suspected TB to be summarized by country. Exact 95% CI to be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Gates MRI, Study Director — Gates Medical Research Institute
Locations (36):
- Investigational Site, Dhaka, Bangladesh
- Brazil (2):
  - Investigational Site, Porto Alegre
  - Investigational Site, Rio de Janeiro
- Investigational Site, Kinshasa, Democratic Republic of the Congo
- Investigational Site, Pune, India
- Indonesia (3):
  - Investigational Site, Bandung, West Java
  - Investigational Site, Bakti
  - Investigational Site, Persabahan
- Kenya (3):
  - Investigational Site, Kisumu
  - Investigational Site, Mombasa
  - Investigational Site, Nairobi
- Mozambique (2):
  - Investigational Site, Manica
  - Investigational Site, Maputo
- Peru (2):
  - Investigational Site, Comas
  - Investigational Site, Lima
- Philippines (5):
  - Investigational Site, Dasmariñas
  - Investigational Site, Iloilo City
  - Investigational Site, Makati City
  - Investigational Site, Mandaluyong
  - Investigational Site, Quezon City
- South Africa (8):
  - Investigational Site, Bloemfontein
  - Investigational Site, Durban
  - Investigational Site, Germiston
  - Investigational Site, Kimberley
  - Investigational Site, Mtubatuba
  - Investigational Site, Soshanguve
  - Investigational Site, Soweto
  - Investigational Site, Three Rivers
- Investigational Site, Banjul, The Gambia
- Uganda (2):
  - Investigational Site, Entebbe
  - Investigational Site, Mulago
- Vietnam (2):
  - Investigational Site, Hà Nội
  - Investigational Site, Ho Chi Minh City
- Zambia (3):
  - Investigational Site, Emmasdale
  - Investigational Site, Lusaka
  - Investigational Site, Ndola

IPD SHARING:
Plan to Share IPD: Yes